CLINICAL TRIAL: NCT01980654
Title: A Multicenter, Open-Label, Phase 2 Study of the Bruton's Tyrosine Kinase (BTK) Inhibitor, Ibrutinib, in Combination With Rituximab in Previously Untreated Subjects With Follicular Lymphoma
Brief Title: Study of Ibrutinib in Combination With Rituximab in Previously Untreated Subjects With Follicular Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pharmacyclics LLC. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PCYC-1125-CA
Record Dates: First submitted 2013-10-24; First posted 2013-11-11 (Estimated); Results first posted 2019-04-16 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-03

CONDITIONS: Follicular Lymphoma; B-cell Lymphoma; Non-Hodgkin's Lymphoma
Keywords: Pharmacyclics (PCYC); PCYC; Lymphoma; Follicular Lymphoma; FL; Rituximab; Ibrutinib; Rituxan; Non-Hodgkin's Lymphoma (NHL); NHL; B-cell Lymphoma
MeSH Terms: conditions — Lymphoma, Follicular; Lymphoma, B-Cell; Lymphoma, Non-Hodgkin; Lymphoma | interventions — ibrutinib; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Main Study Arm 1 (Experimental): Subjects enrolled into this arm will receive ibrutinib continuously until disease progression or unacceptable toxicity. In addition, subjects will receive rituximab once weekly for four doses for the first four weeks of study treatment.
  Interventions: Drug: Ibrutinib; Drug: rituximab
- Exploratory Study Arm 2 (Experimental): Subjects enrolled into this arm will receive ibrutinib continuously as a single agent for the first eight weeks, then ibrutinib concurrently with rituximab once weekly for four doses. After the rituximab treatment, subjects will receive ibrutinib continuously until disease progression or unacceptable toxicity.
  Interventions: Drug: Ibrutinib; Drug: rituximab

INTERVENTIONS:
Drug: Ibrutinib — All subjects will receive 560 mg of Ibrutinib orally.
  Other Names: PCI-32765
Drug: rituximab — All subjects will receive rituximab 375 mg/m2 intravenously
  Other Names: Rituxan

SUMMARY:
This is an open-label, Phase 2 study designed to assess the efficacy and safety of ibrutinib combined with rituximab in previously untreated subjects with Follicular Lymphoma (FL).

DETAILED DESCRIPTION:
This is an open-label, Phase 2 study designed to assess the efficacy and safety of ibrutinib combined with rituximab in previously untreated subjects with FL.

There are two study treatment arms.

Subjects enrolled into main study treatment arm will receive ibrutinib continuously until disease progression or unacceptable toxicity. In addition, subjects will receive rituximab once weekly for four doses for the first four weeks of study treatment.

Subjects enrolled into the exploratory study treatment arm will receive ibrutinib continuously as a single agent for the first eight weeks, then ibrutinib concurrently with rituximab once weekly for four doses. After the rituximab treatment, subjects will receive ibrutinib continuously until disease progression or unacceptable toxicity.

ELIGIBILITY:
Key Inclusion criteria:

1. Histologically documented FL (Grade 1, 2 and 3A)
2. Not previously treated with prior anti-cancer therapy for FL
3. Stage II, III or IV disease
4. At least one measurable lesion ≥ 2 cm in longest diameter by CT and/or MRI scan
5. Men and women ≥ 18 years of age
6. Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2

Key Exclusion criteria:

1. Medically apparent central nervous system lymphoma or leptomeningeal disease
2. FL with evidence of large cell transformation
3. Any prior history of other hematologic malignancy besides FL or myelodysplasia
4. History of other malignancies, except

   1. Malignancy treated with curative intent and with no known active disease present for ≥5 years before the first dose of study drug and felt to be at low risk for recurrence by treating physician.
   2. Adequately treated non-melanoma skin cancer or lentigomaligna without evidence of disease.
   3. Adequately treated carcinoma in situ without evidence of disease.
5. Currently active, clinically significant cardiovascular disease or myocardial infarction within 6 months of screening
6. Known anaphylaxis or Immunoglobulin E (IgE)-mediated hypersensitivity to murine proteins or to any component of rituximab (Rituxan®)
7. Requires anti-coagulation with warfarin or a vitamin K antagonist.
8. Requires treatment with strong cytochrome P450 (CYP) 3A inhibitors.
9. Known bleeding diathesis or hemophilia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2013-12; Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jutta K. Neuenburg, MD, PhD, Study Director — Pharmacyclics LLC.
Locations (12):
- United States (12):
  - Providence Saint Joseph Medical Center, Burbank, California
  - City of Hope, Duarte, California
  - UCLA Medical Center, Los Angeles, California
  - Stanford University, Stanford Care Center, Stanford, California
  - Southeastern Regional Medical Center, Newnan, Georgia
  - Community Health Network Community Regional Cancer Center North, Indianapolis, Indiana
  - Comprehensive Cancer Centers of Nevada, Henderson, Nevada
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Weill Cornell Medical College New York-Presbyterian Hospital, New York, New York
  - Mid-Ohio Oncology/ Hematology Inc, Columbus, Ohio
  - Tennessee Oncology, PLLC The Sarah Cannon Research Institute, Nashville, Tennessee
  - The University of Texas MD Anderson Cancer Center, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Main Study Arm 1 | Exploratory Study Arm 2
Started | 60 | 20
Completed | 60 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Main Study Arm 1 | Exploratory Study Arm 2 | Total
Number analyzed (Participants) | 60 | 20 | 80
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 42 | 12 | 54
  >=65 years | 18 | 8 | 26
Age, Continuous [Median (Full Range); unit: years] | 58.0 [32 to 84] | 55.0 [30 to 75] | 58.0 [30 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 8 | 40
  Male | 28 | 12 | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 6
  Not Hispanic or Latino | 57 | 17 | 74
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 56 | 18 | 74
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 60 | 20 | 80
Baseline B-Symptoms [Count of Participants; unit: Participants] — Criteria used to assess B-symptoms- Subject presenting with at least one of the following:
  Weight loss of >10% for the last 6 months or less; Fever >38C (100.4F) for at least 3 consecutive days within the last 3 months; Drenching night sweats within the last 3 months
  Participants
    B-Symptoms present prior to first dose | 4 | 0 | 4
    B-Symptoms absent | 56 | 20 | 76
Baseline Eastern Cooperative Oncology Group (ECOG) Score [Count of Participants; unit: Participants] — ECOG Performance status = 0 Fully active, able to carry on all predisease performance without restriction. ECOG Performance status = 1 Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, eg, light housework, office work.
  Participants
    Baseline ECOG Score = 0 | 47 | 12 | 59
    Baseline ECOG Score = 1 | 13 | 8 | 21

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR): Proportion of Subjects Achieving the Best Overall Responses of Complete Response (CR) or Partial Response (PR)
Description: Number of subjects achieving the best overall responses of CR or PR prior to the initiation of the next line of antineoplastic therapy as assessed by investigator per the Cheson et al, 2007 criteria. Target lesions are measured by CT, unless MRI is used as the assessment modality for lesions in anatomical locations not amenable to CT. CR is defined as the disappearance of all evidence of disease. PR is defined as >=50% decrease in the sum of the product of the diameters of up to 6 largest dominant masses.
Time Frame: Subjects in Arm 1 will have imaging assessments every 12 weeks for the first 8 assessments, then every 24 weeks. Subjects in Arm 2 will have imaging assessments starting at week 9, then every 12 weeks for 8 assessments, then every 24 weeks.
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study Arm 1 | Exploratory Study Arm 2
Number analyzed (Participants) | 60 | 20
Participants | 51 | 15

2. Secondary Outcome: Duration of Response (DOR)
Description: DOR is defined as the interval between the date of the first documented response (CR, PR) and the date of the first documented evidence of progressive disease (PD) or death. DOR will be analyzed for the subjects who achieve an overall response during the duration of study.
Time Frame: Up to 45 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Main Study Arm 1 | Exploratory Study Arm 2
Number analyzed (Participants) | 51 | 15
months | NA [30.1602 to NA] — The median DOR was not reached so 95% Confidence Interval is not applicable. | NA [24.6078 to NA] — The median DOR was not reached so 95% Confidence Interval is not applicable.

3. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS is defined as the time interval between the date of the first dose and the date of the earliest occurrence of PD or death due to any cause, whichever occurs first. PD is characterized by any new lesion or increase by >=50% of previously involved sites from nadir.
Time Frame: Up to 45 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Main Study Arm 1 | Exploratory Study Arm 2
Number analyzed (Participants) | 60 | 20
months | 41.922 [31.6057 to 41.9220] | NA [23.4908 to NA] — The median PFS was not reached so 95% Confidence Interval is not applicable.

4. Secondary Outcome: Overall Survival (OS)
Description: Subjects will be followed for survival information up to three years after the last dose of study treatment, until new treatment or death, whichever occurs first. OS is defined as the duration of time from the date of the first dose to the date of death from any cause.
Time Frame: Up to 45 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Main Study Arm 1 | Exploratory Study Arm 2
Number analyzed (Participants) | 60 | 20
months | 41.922 [NA to NA] — The 95% Confidence Interval is not applicable because the median OS was estimated based on time to event data. The 95% confidence limit cannot be estimated. | NA [NA to NA] — The median OS was not reached so 95% Confidence Interval is not applicable.

5. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events
Description: Frequency, severity, and relatedness of treatment-emergent adverse events (AEs) Frequency of treatment-emergent AEs requiring discontinuation of study drug or dose reductions
Time Frame: Up to 45 months
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study Arm 1 | Exploratory Study Arm 2
Number analyzed (Participants) | 60 | 20
Participants
  Subjects with any treatment-emergent AE | 60 | 20
  Subjects with any treatment-emergent AE Grade >=3 | 39 | 14
  Subjects with any treatment-related AE | 59 | 20
  Subjects with any treatment-related AE Grade >=3 | 29 | 14
  Subjects with any Ibrutinib-related AE | 57 | 20
  Subjects with any Ibrutinib-related AE Grade >=3 | 29 | 14
  Subjects with any Rituximab-related AE | 50 | 17
  Subjects with any Rituximab-related AE Grade >=3 | 11 | 7
  TEAE leading to ibrutinib dose reduction | 9 | 5
  TEAE Grade >=3 leading to Ibrutinib dose reduction | 6 | 4
  TEAE leading to witholding Rituximab | 1 | 1
  TEAE Grade >=3 leading to witholding Rituximab | 1 | 1
  TEAE leading to discontinuation of Ibrutinib | 14 | 2
  TEAE Grade >=3 leading to discontinuation of Ibrut | 11 | 1
  TEAE leading to discontinuation of Rituximab | 0 | 0
  TEAE Grade >=3 leading to discontinuation of Ritux | 0 | 0
  Subjects with any TE Serious Adverse Event (SAE) | 14 | 6
  Subjects with any TE SAE Grade >=3 | 13 | 5
  Ibrutinib-related SAEs | 6 | 4
  Ibrutinib-related SAEs Grade >=3 | 6 | 4
  Rituximab-related SAEs | 2 | 2
  Rituximab-related SAEs Grade >=3 | 2 | 2

ADVERSE EVENTS:
Time Frame: 3 years, 9 months
Arm/Group | Main Study Arm 1 | Exploratory Study Arm 2
All-Cause Mortality (participants affected / at risk) | 4/60 | 0/20
Serious Adverse Events (participants affected / at risk) | 14/60 | 6/20
Other Adverse Events (participants affected / at risk) | 60/60 | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Main Study Arm 1 (N=60) | Exploratory Study Arm 2 (N=20)
Eosinophilia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 1 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal achalasia (Gastrointestinal disorders) | 1 (2) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 2 (2) | 3 (3)
Death (General disorders) | 2 (2) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 2 (3) | 2 (2)
Urinary tract infection (Infections and infestations) | 1 (2) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Fallopian tube cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cerebral artery stenosis (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (2) | 0 (0)
Vascular encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Main Study Arm 1 (N=60) | Exploratory Study Arm 2 (N=20)
Neutropenia (Blood and lymphatic system disorders) | 9 (11) | 3 (3)
Thrombocytopenia (Blood and lymphatic system disorders) | 8 (13) | 2 (2)
Increased tendency to bruise (Blood and lymphatic system disorders) | 4 (4) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 3 (4) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 5 (5) | 0 (0)
Cardiac flutter (Cardiac disorders) | 1 (1) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Gilbert's syndrome (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 2 (2)
Conductive deafness (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Ear haemorrhage (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 2 (2) | 1 (1)
Dry eye (Eye disorders) | 15 (24) | 4 (7)
Vision blurred (Eye disorders) | 8 (13) | 6 (10)
Lacrimation increased (Eye disorders) | 3 (4) | 6 (8)
Eye irritation (Eye disorders) | 4 (4) | 1 (2)
Eye pruritus (Eye disorders) | 1 (1) | 1 (1)
Diplopia (Eye disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 34 (78) | 12 (30)
Nausea (Gastrointestinal disorders) | 29 (68) | 10 (22)
Constipation (Gastrointestinal disorders) | 16 (32) | 6 (12)
Vomiting (Gastrointestinal disorders) | 16 (30) | 6 (7)
Stomatitis (Gastrointestinal disorders) | 10 (33) | 11 (35)
Abdominal pain (Gastrointestinal disorders) | 12 (13) | 4 (4)
Dyspepsia (Gastrointestinal disorders) | 8 (10) | 3 (3)
Dry mouth (Gastrointestinal disorders) | 4 (4) | 4 (4)
Flatulence (Gastrointestinal disorders) | 5 (5) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 5 (5) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 2 (3) | 3 (3)
Abdominal pain upper (Gastrointestinal disorders) | 4 (6) | 0 (0)
Gingival bleeding (Gastrointestinal disorders) | 4 (6) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 2 (2) | 1 (11)
Abdominal distension (Gastrointestinal disorders) | 2 (2) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 2 (2) | 1 (1)
Chapped lips (Gastrointestinal disorders) | 1 (1) | 1 (1)
Barrett's oesophagus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hypoaesthesia oral (Gastrointestinal disorders) | 0 (0) | 1 (1)
Lip discolouration (Gastrointestinal disorders) | 0 (0) | 1 (1)
Lip ulceration (Gastrointestinal disorders) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (5)
Fatigue (General disorders) | 41 (108) | 15 (30)
Pyrexia (General disorders) | 15 (20) | 4 (5)
Chills (General disorders) | 10 (12) | 1 (1)
Oedema peripheral (General disorders) | 9 (13) | 1 (1)
Peripheral swelling (General disorders) | 5 (7) | 4 (9)
Chest pain (General disorders) | 4 (4) | 2 (2)
Pain (General disorders) | 4 (4) | 2 (2)
Chest discomfort (General disorders) | 4 (4) | 1 (1)
Swelling (General disorders) | 2 (3) | 2 (4)
Malaise (General disorders) | 3 (4) | 0 (0)
Unevaluable event (General disorders) | 0 (0) | 2 (2)
Feeling hot (General disorders) | 0 (0) | 1 (1)
Gait disturbance (General disorders) | 0 (0) | 1 (1)
Generalised oedema (General disorders) | 0 (0) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 3 (5) | 2 (2)
Hepatic function abnormal (Hepatobiliary disorders) | 2 (4) | 1 (7)
Drug hypersensitivity (Immune system disorders) | 3 (3) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 13 (16) | 7 (12)
Urinary tract infection (Infections and infestations) | 13 (28) | 5 (7)
Sinusitis (Infections and infestations) | 7 (8) | 5 (10)
Conjunctivitis (Infections and infestations) | 4 (4) | 1 (1)
Folliculitis (Infections and infestations) | 2 (3) | 2 (2)
Herpes zoster (Infections and infestations) | 4 (5) | 0 (0)
Onychomycosis (Infections and infestations) | 2 (2) | 2 (2)
Tooth infection (Infections and infestations) | 3 (3) | 1 (1)
Cystitis (Infections and infestations) | 0 (0) | 3 (5)
Influenza (Infections and infestations) | 2 (2) | 1 (1)
Oral herpes (Infections and infestations) | 2 (2) | 1 (1)
Pneumonia (Infections and infestations) | 3 (5) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 3 (3) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 2 (2)
Dacryocanaliculitis (Infections and infestations) | 1 (1) | 1 (1)
Ear infection (Infections and infestations) | 1 (1) | 1 (1)
Localised infection (Infections and infestations) | 1 (1) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1) | 1 (1)
Bacterial vaginosis (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Eye infection (Infections and infestations) | 0 (0) | 1 (1)
Prostate infection (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 7 (9) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1)
Streptococcal infection (Infections and infestations) | 0 (0) | 1 (1)
Tinea cruris (Infections and infestations) | 0 (0) | 1 (1)
Tinea pedis (Infections and infestations) | 0 (0) | 1 (1)
Vulvovaginal mycotic infection (Infections and infestations) | 0 (0) | 1 (1)
Wound infection staphylococcal (Infections and infestations) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 14 (16) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 5 (8) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 3 (4) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Arthropod sting (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 4 (4) | 1 (2)
Alanine aminotransferase increased (Investigations) | 3 (4) | 1 (3)
Blood bilirubin increased (Investigations) | 1 (1) | 1 (2)
Blood pressure increased (Investigations) | 0 (0) | 1 (1)
Low density lipoprotein increased (Investigations) | 0 (0) | 1 (1)
White blood cell count increased (Investigations) | 0 (0) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 6 (7) | 4 (4)
Decreased appetite (Metabolism and nutrition disorders) | 7 (9) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 5 (5) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Abnormal loss of weight (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Polydipsia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 20 (38) | 9 (20)
Arthralgia (Musculoskeletal and connective tissue disorders) | 20 (27) | 3 (5)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 16 (22) | 5 (8)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 (13) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (10) | 2 (3)
Joint swelling (Musculoskeletal and connective tissue disorders) | 4 (8) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 3 (5) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (2)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Headache (Nervous system disorders) | 19 (27) | 5 (10)
Dizziness (Nervous system disorders) | 13 (18) | 9 (19)
Paraesthesia (Nervous system disorders) | 9 (20) | 8 (19)
Memory impairment (Nervous system disorders) | 9 (13) | 5 (9)
Hypoaesthesia (Nervous system disorders) | 3 (3) | 1 (2)
Cognitive disorder (Nervous system disorders) | 3 (3) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 3 (4) | 0 (0)
Tremor (Nervous system disorders) | 2 (2) | 1 (1)
Migraine (Nervous system disorders) | 1 (1) | 1 (1)
Restless legs syndrome (Nervous system disorders) | 1 (1) | 1 (1)
Dyskinesia (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 9 (9) | 0 (0)
Insomnia (Psychiatric disorders) | 8 (10) | 1 (1)
Depression (Psychiatric disorders) | 3 (3) | 0 (0)
Haematuria (Renal and urinary disorders) | 4 (4) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 2 (2) | 2 (2)
Dysuria (Renal and urinary disorders) | 1 (2) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Nocturia (Renal and urinary disorders) | 0 (0) | 1 (1)
Polyuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Vulvovaginal dryness (Reproductive system and breast disorders) | 0 (0) | 2 (2)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Dyspareunia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vulvovaginal erythema (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vulvovaginal pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 20 (26) | 6 (9)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 12 (23) | 4 (8)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 10 (11) | 5 (6)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 5 (9) | 2 (4)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6 (9) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 2 (2)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 18 (32) | 8 (10)
Dry skin (Skin and subcutaneous tissue disorders) | 7 (7) | 3 (3)
Onychoclasis (Skin and subcutaneous tissue disorders) | 8 (9) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 7 (12) | 2 (2)
Rash erythematous (Skin and subcutaneous tissue disorders) | 7 (9) | 1 (1)
Petechiae (Skin and subcutaneous tissue disorders) | 6 (13) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 4 (6) | 1 (1)
Nail disorder (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (3) | 2 (3)
Skin fissures (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 2 (3) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 2 (3) | 1 (1)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Rash macular (Skin and subcutaneous tissue disorders) | 2 (3) | 1 (2)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (2)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Rosacea (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Eczema nummular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Exfoliative rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Koilonychia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Nail discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pyoderma gangrenosum (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Scab (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 10 (12) | 2 (3)
Hot flush (Vascular disorders) | 4 (4) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2016-09-12): https://cdn.clinicaltrials.gov/large-docs/54/NCT01980654/Prot_000.pdf
  • Statistical Analysis Plan (2017-10-27): https://cdn.clinicaltrials.gov/large-docs/54/NCT01980654/SAP_001.pdf